CLINICAL TRIAL: NCT06478628
Title: Insomnia in Patients Participating in Interdisciplinary Pain Rehabilitation
Status: Enrolling by invitation | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Unicare (Unknown)
Responsible Party: Sponsor
Other Study IDs: 547864
Record Dates: First submitted 2024-06-24; First posted 2024-06-27 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Musculoskeletal Pain; Insomnia
MeSH Terms: conditions — Musculoskeletal Pain; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Unicare Helsefort: Patients taking part in rehabilitation due to pain at Unicare Helsefort
  Interventions: Behavioral: Inpatient rehabilitation
- Unicare Hokksund: Patients taking part in rehabilitation due to pain at Unicare Hokksund
  Interventions: Behavioral: Inpatient rehabilitation; Behavioral: Outpatient day rehabilitation
- Unicare Coperio: Patients taking part in rehabilitation due to pain at Unicare Coperio
  Interventions: Behavioral: Outpatient day rehabilitation
- Unicare Jeløy: Patients taking part in rehabilitation due to pain at Unicare Jeløy
  Interventions: Behavioral: Inpatient rehabilitation; Behavioral: Outpatient day rehabilitation
- Unicare Friskvern: Patients taking part in rehabilitation due to pain at Unicare Friskvern
  Interventions: Behavioral: Outpatient day rehabilitation

INTERVENTIONS:
Behavioral: Inpatient rehabilitation — Inpatient multimodal rehabilitation in specialist health care
  Groups: Unicare Helsefort; Unicare Hokksund; Unicare Jeløy
Behavioral: Outpatient day rehabilitation — Multimodal rehabilitation in specialist health care with program lasting whole work days
  Groups: Unicare Coperio; Unicare Friskvern; Unicare Hokksund; Unicare Jeløy

SUMMARY:
The main purpose of this project is to conduct a prospective cohort study in order to better understand the importance of insomnia symptoms in patients referred to interdisciplinary rehabilitation due to chronic pain. Moreover, this project will also raise awareness on how insomnia symptoms, alone, and in interplay with factors such as function, psychological distress, physical activity, and fatigue impact on patient's prognosis and work ability. Our aim is that this knowledge can be used to design new interventions and improve rehabilitation programs for this patient group.

DETAILED DESCRIPTION:
Insomnia is a vast problem among patients with chronic musculoskeletal pain. Despite the close relation between pain and sleep, sleep quality has received little attention in rehabilitation programs for patients with pain. So far, there is a lack of studies investigating the association between insomnia and chronic pain in patients referred to interdisciplinary rehabilitation. Identifying subgroups of the population with higher burden of poor sleep will aid clinicians to tailor treatment and prevention strategies. Moreover, knowledge on how insomnia symptoms fluctuate throughout the rehabilitation program and how insomnia symptoms interact with factors such as mental distress, physical activity, and fatigue impact on patient's recovery (e.g., the prognosis of pain, quality of life, and work participation) can be used to develop and implement more successful rehabilitation programs.

This is a cohort study primarily designed to address sleep problems in patients referred for pain rehabilitation by using questionnaire data from the rehabilitation centers linked to registry data. This study will constitute both a cross-sectional survey among patients referred to rehabilitation before they participate in rehabilitation. In addition to questionnaires, administrative data and clinical data, these data will be linked to national health registries on prescriptions, health care use and sickness absence. Potential participants are patients referred to rehabilitation at five different Unicare rehabilitation centers in Norway (Unicare Helsefort, Unicare Coperio, Unicare Hokksund, Unicare Friskvern and Unicare Jeløy) due to long-term pain complaints.

ELIGIBILITY:
Inclusion Criteria:

* Take part in rehabilitation for long-term pain complaints at one of the five centers
* Consented to research

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential participants are patients referred to rehabilitation at five different Unicare rehabilitation centers in Norway (Unicare Helsefort, Unicare Coperio, Unicare Hokksund, Unicare Friskvern and Unicare Jeløy) due to long-term pain complaints. Potential participants are referred to outpatient or inpatient rehabilitation or a shorter assessment stay (where the goal is to assess what is the best treatment option for the patient). Referrals to the rehabilitation centers are done by the patients' general practitioner or by specialist healthcare. All referrals are considered at the regional unit for referrals (Regionalt henvisningsmottatak) in mid- or southeast Norway who judge whether they fulfill the criteria for rehabilitation in specialist health care.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Insomnia | Baseline
  Measured by Insomnia severity index (ISI)
Pain intensity | Baseline
  Measured by visual analogue scale (0 to 100 scale)

SECONDARY OUTCOMES:
Health-related quality of life | Baseline
  Measured by the the 5-level EQ-5D version (EQ-5D-5L) questionnaire. The index value range ranges from -0.285 to 1, where lower values indicate poorer health-related quality of life.
Fatigue | Baseline
  Measured using a visual analogue scale from 0 to 100
Function | Baseline
  Measured by the patient-specific functional scale (PSFS)
Physical activity | Baseline
  Measured by questions from the HUNT study
Workability | Baseline
  Measured by the workability index single item (self- assessed work ability on a 0-10 scale)
Symptoms of anxiety and depression | Baseline
  Measured by the Hopkins Symptom Checklist-25 (HSCL-25), mean score calculated (1-4)
Prescriptions | Up to five years before rehabilitation and one year after rehabilitation
  Use of sleep psychotropic medications, and pain medications based on registry data
Sickness absence | Up to five years before rehabilitation and one year after rehabilitation
  Use of medical benefits based on registry data
Health care use | Up to five years before rehabilitation and one year after rehabilitation
  Health care use in primary care based on registry data

CONTACTS AND LOCATIONS:
Overall Officials: Solveig K. Grudt, Msc, Study Chair — National Taiwan Normal University
Locations (1):
- Unicare Helsefort, Rissa, Norway